CLINICAL TRIAL: NCT03952715
Title: Can Training Increase Reporting Accuracy and Study Power in Human Pain Trials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 016/18
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Healthy; Placebo Response
Keywords: Focus analgesia selection test (FAST); Experimental pain variability; Placebo effect; Evoked pain training (EPT)
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evoked pain training (Experimental)
  Interventions: Drug: Ibuprofen 400 mg; Drug: Placebo oral tablet
- Control (Experimental)
  Interventions: Drug: Ibuprofen 400 mg; Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Ibuprofen 400 mg — Each subject will receive Ibuprofen once, in between two psycho-physical assessments. Between the drug intake and the second assessment the subject will have to wait for 40 minutes.
Drug: Placebo oral tablet — Each subject will receive Placebo (sugar pill) once, in between two psycho-physical assessments. Between the placebo pill intake and the second assessment the subject will have to wait for 40 minutes.

SUMMARY:
In previous studies, results of both the Focused Analgesia Selection Test (FAST) procedure, a method to assess pain-reporting accuracy, and the Evoked Pain Training (EPT) procedure, aimed to improve pain-reporting accuracy, correlated with the placebo response. The objectives of the current project were to determine if EPT (1) increases pain reporting accuracy and (2) affect the placebo response in experimental pain study.

DETAILED DESCRIPTION:
Analgesic trials suffer from low assay-sensitivity, and experts in the field are concerned that many previous negative analgesic trails might be regarded as failed trails. Major contributor to this concern is the large placebo response observed in analgesic clinical trials. Recent findings from the investigators group suggest that improving pain reporting accuracy could increase analgesic trials assay sensitivity by reducing the placebo response. In previous studies, the investigators developed the Focused Analgesia Selection Test (FAST), a method to assess pain reporting accuracy. Later on, the investigators developed the Evoked Pain Training (EPT), aimed to improve pain reporting accuracy. Both these methods constitute the core of this project. The objectives of the current project are to determine if subject training increases (1) pain reporting accuracy and (2) the power of an analgesic trial.

Summary of main methods This project objectives will be achieved by preforming a two-stage study. First, all subjects undergo baseline assessments, including assessment of pain reporting accuracy (the FAST procedure) (visit #1). Then, subjects enter the first study stage (training stage), in which half of study subjects (n=50) undergo training to improve pain reporting accuracy. The training comprise of three in-clinic visits (visits #2, 3, 4) in which subjects receive feedback on accuracy of pain reports in response to noxious stimuli of various intensities (the EPT procedure). The EPT is based on repeated application of the FAST procedure, while providing feedback to subjects in between applications. The other half of subjects (n=50) undergo a "shame-training". After completion of the training phase, all subjects enter an experimental cross-over study design (second study phase) comprised of two in-clinic visits (visits 5 and 6). In each of these two visits, subjects undergo a battery of experimental pain tests (pre-treatment assessment), take one of two pills (either Ibuprofen 400 mg or identical sugar pill) in a random order, wait approximately 1 hour, and then undergo the same pain tests again (post-treatment assessment).

ELIGIBILITY:
Inclusion Criteria:

* Absence of neurological, psychiatric, or chronic pain disorders.
* Have used at list once Ibuprofen, and not sensitive to NSAIDs.
* Ability to give informed consent, communicate, and understand the purpose and instructions of this study.

Exclusion Criteria:

* Presence of diagnosed psychiatric disorders, cognitive and /or neurological deficits.
* Use of analgesic, anti-depressant or anti-enxiayoltic medications on a regular basis (except for oral contraceptives).
* Pregnancy.
* Never used NSAIDs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Pain reporting accuracy | Fast procedure itself (49 heat stimuli, from 7 designated heat temperatures, given in a random block-order design) lasting approximately 20 minutes.
  Subjects will be asked to report their pain on numerical pain scale (NPS) ranging from 0, denoting "no pain", to 10, denoting "the worst pain imaginable".
Change in experimental pain perception due to drug/placebo pill intake | Mechanical and thermal stimuli before the drug/placebo (Pre-drug/placebo) until receiving the same stimuli 40 minutes after taking the drug/placebo pill (Post-drug/placebo).
  Subjects will be asked to report their pain on numerical pain scale (NPS) ranging from 0, denoting "no pain", to 10, denoting "the worst pain imaginable". The placebo effect (Δ) will be calculated as the difference between the mean NPS.

SECONDARY OUTCOMES:
Evoked pain training | Fast procedure itself (49 heat stimuli, from 7 designated heat temperatures, given in a random block-order design) lasting approximately 20 minutes. There are 3 training visits, each training consists of 2 FAST procedure and last approximately 1 hour.
  Subjects will be asked to report their pain on numerical pain scale (NPS) ranging from 0, denoting "no pain", to 10, denoting "the worst pain imaginable".

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, The Clinical Pain Innovation Lab, Haifa, Israel